CLINICAL TRIAL: NCT04238793
Title: A Phase 1/2a, First-in-Human, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Therapeutic Activity of Single Ascending Doses of KLS-2031 Administered by Transforaminal Epidural Injection in Patients With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Single Ascending Doses Study of KLS-2031 in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS-GIG-001-01
Record Dates: First submitted 2019-12-24; First posted 2020-01-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Neuropathic Pain From Lumbosacral Radiculopathy
Keywords: Neuropathic pain from lumbosacral radiculopathy; Lumbosacral radiculopathy; LSR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Dose 1 (low dose: 1×1011 VG/500 μL solution) or Placebo
  Interventions: Drug: KLS-2031; Other: Placebo
- Cohort 2 (Experimental): Dose 2 (medium dose: 1×1012 VG/500 μL solution) or Placebo
  Interventions: Drug: KLS-2031; Other: Placebo
- Cohort 3 (Experimental): Dose 3 (high dose: 1×1013 VG/500 μL solution) or Placebo
  Interventions: Drug: KLS-2031; Other: Placebo

INTERVENTIONS:
Drug: KLS-2031 — KLS-2031 administered by transforaminal epidural injection
Other: Placebo — Normal Saline (0.9%) administered by transforaminal epidural injection

SUMMARY:
Escalating single-dose design study to determine the safety, tolerability, and analgesic activity of KLS-2031

DETAILED DESCRIPTION:
This is a first-in-human (FIH), multicenter, double-blind, placebo-controlled, parallel-group, escalating single-dose design study to determine the safety, tolerability, and analgesic activity of KLS-2031 administered by transforaminal epidural injection to subjects aged 18 to 75 years with neuropathic pain due to LSR.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, subjects must have met the following criteria at Visit 1 (Screening,

Day -56 to Day -15):

1. The subject signed a written informed consent for study participation including the 1-year double-blind treatment period and 1-year, open-label, long-term extension period.

   Informed consent must have been obtained before any screening activities are conducted.
2. The subject, male or female, must have been between the ages of 18 and 75 years, inclusive.
3. The subject must have had a body mass index of ≤35 kg/m².
4. The subject must have had a diagnosis of pain due to LSR, with all of the following characteristics:

   1. The subject perceived pain in 1 or both lower limbs at areas that are consistent with the area innervated by the lumbar 4 or 5 or sacral 1 (L4, L5, S1) nerve roots, with or without other sensory symptoms in the affected areas (typically, the pain may have been perceived in the buttock, thigh, calf, leg, foot, or toes). If both limbs were affected, pain had to be asymmetrical (ie, pain worse in 1 limb).
   2. Pain in the leg radiated to below the knee.
   3. Pain in the leg was worse during rest and/or at night and not solely present upon walking.
   4. The history of the pain suggested that the cause of the LSR was due to the injury of the lumbosacral nerve root(s) by degenerative disease of the vertebrae in the lumbosacral spine or associated soft tissues (including the intervertebral discs).
   5. The duration of the pain since onset was ≥6 months.
   6. Based on clinical history, the intensity of the neuropathic (leg) pain had been stable during the 4-week period before screening (the pain may have fluctuated and may have been worse at night or at rest but was present on most days of the week).
5. Pain in the leg (worse affected leg) was worse than pain in the back.

Exclusion Criteria:Subjects were excluded from the study if 1 or more of the following criteria were applicable:

1. The subject had:

   1. Neuropathic pain due to causes other than that specified in the inclusion criteria (eg, postherpetic neuralgia; painful diabetic neuropathy; mononeuritis multiplex; central poststroke pain; spinal abscess, infection, hematoma, spondylolisthesis with displacement, or malignancy; phantom limb pain; peripheral neuropathy due to alcoholism, malignancy, HIV, syphilis; drug abuse; vitamin B12 deficiency; hypothyroidism; liver disease; toxic exposure).
   2. Radicular pain at more than 1 spinal level, unstable spine, spondylolisthesis (>Grade 1), spondylolysis, caudal equina syndrome, arachnoiditis, progressive neurological deficit, moderate to severe central spinal canal stenosis (congenital or acquired) from other origins, vertebral compression fracture(s).
   3. Pain that was associated with a substantial somatic pain component in lower limbs or other parts of the body apart from the back (eg, non-neuropathic/musculoskeletal pain) or more than 1 cause or potential cause for pain symptoms in low limbs.
   4. Any painful concurrent rheumatic disease such as, but not limited to, fibromyalgia, rheumatoid arthritis, or osteoarthritis that in the investigator's opinion would have prevented the subject from reliably delineating or assessing his/her pain due to LSR. Note: Any question regarding the acceptability of the etiology of the neuropathic pain was to be discussed with the medical monitor.
2. Had lumbar stenosis with pain present solely upon walking. Presence of lumbar narrowing on MRI was acceptable if the pain was not solely present upon walking.
3. In the investigator's opinion, the subject was unable to reliably delineate or assess his/her own pain by anatomical location/distribution (eg, the subject could not reliably tell the difference between his/her back pain and lower limb pain and could not rate the intensity of each separately).
4. The subject had pain in the lower limbs solely upon walking and not at rest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of KLS-2031 | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52
  Frequency and nature of AEs, laboratory test results, vital sign measurements, physical and complete neurological examinations, and 12-lead electrocardiograms (ECGs)

SECONDARY OUTCOMES:
Long-term safety and tolerability of KLS-2031 | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 78, Week 104
  Frequency and nature of AEs, laboratory test results, vital sign measurements, physical and complete neurological examinations, and 12-lead ECGs
Local safety and tolerability (including AEs, clinical laboratory parameters, and physical examination) of administration by transforaminal epidural injectionepidural injection as measured by the occurrence of injection site reactions | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52
  The occurrence of injection site reactions
Change from baseline in weekly mean of the average daily pain score | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
  calculated as the average of the subject's last 4 available PI-NRS daily scores in the week before the study visit
Change from baseline in Galer Neuropathic Pain Scale (Galer NPS) | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Number and percentage of subjects who have ≥30% and ≥50% reduction from baseline in the average daily pain score (PI-NRS) | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Time (number of weeks) to ≥30% and ≥ 50% reduction from baseline in the average daily pain score (PI-NRS) | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Number and percentage of subjects who are much improved or very much improved from baseline | Week 12, Week 26, Week 52, Week 104
  based on the Patient Global Impression of Change (PGIC)
Change from baseline in the modified Modified Roland-Morris Disability Questionnaire (RMDQ) scores (back pain and leg pain) | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Amount of rescue medication used (in terms of dosage/day) | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52
Time to treatment failure | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52
  , defined as the day and time a subject starts pain medication other than acetaminophen for the treatment of neuropathic pain
Change from baseline in the Simple Profile of Moods States (POMS) - 2 Short Form total score and domain scores | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Change from baseline in Daily Sleep Interference Scale (DSIS) score | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52, Week 104
Change from baseline in the Short Form-36 v2 (SF-36v2) score | Week 12, Week 26, Week 52, Week 104
Assessment of suicidality | Week 1, Week 2, Week 4, Week 12, Week 26, Week 52
  using the Columbia Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- Kolon Investigative Site : CenExel JBR, Salt Lake City, Utah, United States